CLINICAL TRIAL: NCT06219798
Title: Evaluation of a Multidisciplinary Care Pathway on the Evolution of Renal Function in Patients With Advanced Chronic Kidney Disease
Brief Title: Evaluation of a Pathway on the Evolution of Renal Function in Patients With Advanced Chronic Kidney Disease
Acronym: EPSER
Status: Recruiting | Type: Observational
Sponsor: Association d' Utilisation du Rein Artificiel SANTE (Other)
Responsible Party: Principal Investigator, PAGES Helene, Principal Investigator, Association d' Utilisation du Rein Artificiel SANTE
Other Study IDs: Pathway CKD 4 and 5
Record Dates: First submitted 2023-11-20; First posted 2024-01-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Kidney Function Issue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Name of Arm 1: Study group: Description: Full participation (medical + dietitian+ specialist nurse)
  Interventions: Diagnostic Test: GFR
- Name of Arm 2: Control 1: Description: Partial participation (medical+ dietitian OR specialist nurse)
  Interventions: Diagnostic Test: GFR
- Name of Arm 3: Control 2: Description: No participation (medical visit only)
  Interventions: Diagnostic Test: GFR

INTERVENTIONS:
Diagnostic Test: GFR — Exit of the study due to death, dialysis, or transplantation
  Other Names: Renal outcome

SUMMARY:
The number of incident and prevalent patients with end stage renal disease on dialysis treatment is increasing in France and worldwide. A quarter of dialysis patients are initiating dialysis urgently through central venous catheters and the number of patients registered in the waiting list for renal transplantation before dialysis initiation is very low. This is also reflected in the very low number of pre-emptive renal transplantations.

In order to reduce the number of dialysis patients, the French state has induced a national program proposing a multidisciplinary care pathway including the nephrology visits and at least one consultation with a dietitian and a specialist renal nurse in all patients with Chronic Kidney Disease stage 4 and 5.

The aim of this single-center retrospective study is to evaluate the influence of the complete, partial or no participation in this program on the evolution of renal function and clinicobiological parameters in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* All stage 4 and 5 Chronic Kidney Disease patients that were included in the program from 01/01/2021 to 31/12/2021 in the clinics of AURA SANTE

Exclusion Criteria:

* Patients without a medical follow up during this year (2021)
* Patients with insufficient or no data during the 24 month of follow up period
* Active treatment with corticosteroids, cytotoxic or immunosuppressive drugs, ongoing infection, autoimmune disease or active tumor process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 4 and 5 Chronic Kidney Disease patients that were included in the program from 01/01/2021 to 31/12/2021 in the clinics of AURA SANTE
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate | Every 6 months for 24 months
  The estimated Glomerular filtration rate is estimated with the CKD-EPI formula adjusted for 1.73m2 of body surface area and produced in ml/min/1.73m2 of body surface area

SECONDARY OUTCOMES:
Patients survival rate | Every 6 months for 24 months
  Number of deaths during the sudy period
Renal survival rate | Every 6 months for 24 months
  Number of patients initiating dialysis during the study period
Haemoglobin levels | Every 6 months for 24 months
  Evolution of haemoglobin levels during the study period in gram/dL
Plasma Calcium levels | Every 6 months for 24 months
  Evolution of plasma calcium levels during the study period in mg/dL
Plasma Phosphate levels | Every 6 months for 24 months
  Evolution of plasma phosphate levels during the study period in mg/dL
Plasma parathyroid hormone levels | Every 6 months for 24 months
  Evolution of plasma parathyroid hormone levels during the study period in pg/ml
Plasma alcaline reserve levels | Every 6 months for 24 months
  Evolution of plasma alcaline reserve levels during the study period in mmol/l
24h salt consumption | Every 6 months for 24 months
  Evolution of salt consumption during the study period in g/24h
24h protein consumption | Every 6 months for 24 months
  Evolution of protein consumption during the study period in g/24h
Quality of life score | through study completion, an average of 6 months
  Scores from Evaluation Quality of life,5 dimensions, 5 levels (EQ-5D-5L), the higher the score the better the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Aura Sante, Chamalières, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
The chief investigator is going solely to include and analyse data without sharing them with anybody else